CLINICAL TRIAL: NCT02247635
Title: Development of a Methodology for Diagnosis and Promoting Adherence to Treatment of Patients With Chronic Diseases and Evaluation of Their Impact on Cardiovascular Risk Factors
Brief Title: Effect of a Treatment of Lifestyle Changes on the Prevalence of Metabolic Syndrome and Body Weight in Mexican Women
Acronym: MPATPCDNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mexican National Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Simon Barquera, MD, MS, PhD, Director of Research in Nutrition Policy and Programs., Mexican National Institute of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINYS 410; 000000000044415 (Other: Council of Science and Technology)
Record Dates: First submitted 2014-09-17; First posted 2014-09-25 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Obesity; Diabetes; High Blood Pressure; Dyslipidemia
Keywords: Treatment adherence; Behavioral model of health care; Healthy lifestyle; Chronic metabolic diseases; Metabolic syndrome; Obesity
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Hypertension; Dyslipidemias; Treatment Adherence and Compliance; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional medical treatment (No Intervention): Based on the clinical guidelines of the Ministry of Health, medical treatment was provided and consisted in counseling for chronic diseases such as obesity, hyperglycemia, hypertension, dyslipidemia
- Healthy lifestyle and adherence (Active Comparator): 1) Maintain a caloric restriction of 500kcal in overweight adults, 2) Have a total fat intake <30% (including cholesterol and trans fat), 3) A total intake of complex carbohydrates for 50%, 3) 30g fiber, 4) Perform at least 30 minutes of moderate physical activity at least 5 days a week; 5) Maintain education and behavioral therapy changes in your lifestyle.
  Interventions: Behavioral: Healthy lifestyle and adherence

INTERVENTIONS:
Behavioral: Healthy lifestyle and adherence — Behavioral intervention to improve adherence to treatment and 1) Maintain a caloric restriction of 500kcal in overweight adults, 2) Have a total fat intake <30% (including cholesterol and trans fat), 3) A total intake of complex carbohydrates for 50%, 3) 30g fiber, 4) Perform at least 30 minutes of moderate physical activity at least 5 days a week; 5) Maintain education and behavioral therapy changes in your lifestyle.
  The model consists of monthly visits to the doctor, nutritionist and psychologist, for screening cardiometabolic risk factors, to know limitations on treatment adherence, to start intervention to evaluate reasons for success or failure, to evaluate and maintain motivation to adherence to diet, physical activity and medication and long-term care
  Arms: Healthy lifestyle and adherence

SUMMARY:
The metabolic syndrome is a group of cardiometabolic risk factors that reflect a sedentary lifestyle and the excessive intake of food among the risk factors that comprise it are located the obesity, hyperglycemia, dyslipidemia and hypertension.

It has been observed that the interventions of lifestyle changes that promote weight loss through the practice of physical activity and intake of a hypocaloric diet, reduce the prevalence of chronic diseases such as Metabolic syndrome.

Adherence is defined as the extent to which a person's behaviour - taking medication, following a diet, and/or executing lifestyle changes, corresponds with agreed recommendations from a health care provider. The World Health Organization has estimated that in developing countries, as in Mexico, less than 27% of people with chronic diseases will continue treatment as directed.

Adherence to treatment of chronic disease is a multifactorial problem that includes not only patient-related barriers, but also providers of health services and social security systems themselves. Furthermore, as WHO has pointed out, as increasing prevalence of chronic non-adherence to treatment will become a global problem even more serious.

The purpose of this study is develop and implement a methodology to overcome barriers affecting adherence to treatment of women over 20 years with non-communicable diseases such as metabolic syndrome (diabetes , hypertension and dyslipidemia) evaluating its impact through various quantitative indicators such as weight loss or metabolic syndrome prevalence.

This study will include two phases:

1. Phase 1. Design. Qualitative methodology was used primarily to identify the barriers faced by individuals to adhere to treatment. From this methodology, we developed a tool to assess adherence to treatment of subjects with these conditions and then an intervention to improve it.
2. Phase 2. Implementation of intervention (24 weeks). To recruite a group of 180 overweight and two of the following comorbidities: diabetes mellitus, dyslipidemia or hypertension. All study subjects will be randomized to a control group and intervention. The control group will receive a medical traditional clinical care. The intervention group will receive a lifestyle treatment with behavioral intervention to improve adherence for improve eating behaviors, physical activity and metabolic control.

DETAILED DESCRIPTION:
The World Health Organization estimates that worldwide one billion adults are overweight. In Mexico, the prevalence of overweight and obesity using data from 2006 was nearly 70% in men and women over 20 years.

Being overweight is associated with other co-morbidities such as diabetes mellitus (79.4%), hypertension (78.0%) and dyslipidemia (82.8%). WHO has estimated that over 50% of these patients have a poor grip and do not follow their treatment as indicated, generating costs for managing these diseases of until $ 100 billion each year. Improve the effectiveness of interventions on adherence to treatment, will significantly improve the health of these patients and help reduce costs involving health systems.

The obesity and comorbidities affect 41% of the adults in Mexico and increases up to five times the risk of developing cardiovascular disease and type 2 diabetes and up to three times the risk of developing coronary artery disease and myocardial infarction. Therefore, these diseases are currently one of the main problems of public health in Mexico.

Adherence to short and long term is the result of a complex process that develops through different stages: the acceptance of diagnosis, the perceived need for treatment successfully, motivation, and skills training available, the ability to overcome the barriers or difficulties arise, and maintenance of achievements over time.

The lack of adherence to chronic disease is a multifactorial problem that includes not only patient-related barriers, but also with service providers and health systems. Poor adherence to long-term therapies severely compromises the effectiveness of treatment and negatively impacts the quality of life of patients.

It has been observed that the interventions of lifestyle changes that promote weight loss through the practice of physical activity and intake of a hypocaloric diet, reduce the prevalence of Metabolic diseases and achieve a better control.

The changes in lifestyle are the foundation of any strategy for the treatment of chronical diseases . The patients require counseling to effect change in their behavior and improve their risk of mortality and morbidities. So far, interventions to improve treatment of patients with chronic diseases, not including diet and exercise recommendations, has not reported any significant positive change. Moreover, in Mexico there is still no method or reference tool to assess adherence. It has been reported that healthy lifestyles achieve positive changes on cardiovascular risk factors, however, no known methodology to help patients overcome the barriers that prevent them from adopting and adhering to the recommendations that are prescribed providers of health services. Therefore, the objective of this study is to assess if a multidisciplinary treatment that stimulates the constant practice of physical activity and intake of a hypocaloric diet, reduces the prevalence of metabolic chronic diseases such as obesity, diabetes, hypertension and dyslipidemia, and improves the control, in comparison with a traditional medical treatment in Mexican women. Also, to develop a methodology validated in Mexican population to identify barriers that affect adherence to treatment assessing their impact through a variety of quantitative indicators of health.

This project was conducted in 2 phases.

PHASE 1 Development of the tool for identifying barriers. In a private hospital care to chronic noncommunicable diseases, were called patients with co-morbidities associated with overweight and obesity (diabetes mellitus, dyslipidemia, hypertension) to identify common barriers they face to adequately follow through treatment the application of a validated questionnaire. The results will be used as reference for the discussion of traditional treatment algorithms based on the Mexican standards for the management of obesity, hypertension, diabetes and dyslipidemia.

PHASE 2. Design and implementation of the intervention

Phase 2 began with the recruitment of study subjects. The recruitment was done by a local advertising campaign that included posters and leaflets in the city the Cuernavaca, Morelos. México.

Were recruited a group of 180 patients with overweight and two of the following co-morbidities: diabetes mellitus, dyslipidemia or hypertension. All study subjects will be randomized to a control group and intervention. The intervention will last 24 weeks. The control group will receive traditional clinical care and the intervention group will receive a behavioral intervention to improve adherence.

The design of the intervention is based in the the stages-of-change model (also referred to as the transtheoretical model) identifies five stages through which individuals progress as they change behaviours, and stage-matched strategies that predict progress to each subsequent stage of change.

The stages of change are:

Precontemplation at this stage the subject does not plan to make an effort to adhere to treatment or to change your behavior. (Not considering changing behavior in the next 6 months),

The second is called "contemplation", the person admits that there is a risk behavior or beneficial and begin thinking about trying to change or adopt. (Considering changing behavior in the next 6 months),

The third is "preparation" in this stage the person intends to initiate behavior change, strategies and plans to acquire solutions. (Planning to change behavior during the next 30 days),

The fourth is "action" has become the person intended in the expected action (in this study the action is to improve adherence to treatment). (Currently changing behavior)

The fifth is "maintenance", here the change has been established as usual. (Successful behavior change for at least 6 months).

There is a sixth stage called "relapse", where the person returns to the behaviors that had been changed, abandoned the effort and go to the pre-action stages.

Stages of change describe an individual's motivational readiness to change.

The specific tools that contain the intervention program are:

Preparation

At this stage various strategies will be developed:

* Educational texts
* Individual medical advice
* Written contract of engagement The objective of this stage is to make the individual reflect on his health.

Action At this stage the individual begins proper actions to get a better adherence It will provide enough printed material that allows it to achieve its goals in diet, physical activity and taking medications.

There will be a computerized database (software) with which you can update the progress and barriers presented by the individual and be able to access either the nutritionist doctor or psychologist

Description of the tools:

* Educational texts. Based on feedback from patients and doctors, nutritionists and psychologists experts, will be designed brochures and educational leaflets with practical advice to achieve intermediate goals and the end of each treatment.
* Consultation and personalized feedback Develop a scheme for service providers (doctors, nutritionists and psychologists) to provide attention individual, the query will be adjusted to the level of adherence achieved.

In the query are used as reference treatment guidelines of the ADA and the Third Adult Treatment Panel (ATP III).

* Nutrition. The consultation will be given by a nutritionist trained to give dietary treatment based on available activities and times of the patient.
* Physical activity. The type of activity will be designed by an expert in the field and will be prescribed by nutritionist taking into account the patient's age and abilities.

Data collection will be done with different tools according to the phase of the project

Phase 1:

a) Identification of barriers to treatment through the application of validated questionnaires.

Phase 2:

1. Identification and socioeconomic data through the application of two questionnaires.
2. Anthropometry: weight with scale Tanita model BC-418. Height with stadiometer SECA, model 220. Waist with a ribbon of flexible glass fiber of 0.5 cm in width and a precision of 1 mm.
3. The measurement of intima-media thickness of carotid is made with Ultrasound SONOSITE PLUS model 180.
4. Collection of biological samples for determination of biochemical parameters like glucose, glycosylated hemoglobin, total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides.

Variables

Dependent. The dependent variable or outcome will be reduction in the prevalence of obesity and comorbidities (such as hypertension, diabetes, dyslipidemia), and control measured through weight loss, and decrease in blood pressure, fasting glucose, and cholesterol.

Independent. The independent variable is the lifestyle and behavioral program.

Data Analysis. Will present descriptive statistics for the dependent variables weight, fasting glucose, HbA1c, triglycerides, HDL-C, LDL-C, blood pressure and intima-media thickness.

Each group will analyze the mean difference in measurement time (initial, intermediate and final) for mean difference test

The differences between the control and intervention group were analyzed using three strategies: 1) by intention to treat (including patients who dropped out), 2) full support to the intervention (patients who completed the program), and 3) for proper administration of the intervention, ie an analysis will be specific to those subjects who received the intervention effectively by the physician and nutritionist (patients intervened correctly).

ELIGIBILITY:
Inclusion Criteria:

* Women from 19 to 65 years old
* Body mass index ≥ 25.0 - ≤39.9 or abdominal obesity
* With previous medical diagnosis:

  1. high fasting glucose
  2. high blood pressure
  3. dyslipidemia.

Exclusion Criteria:

* Currently pregnant or breast-feeding.
* Anxiety and depression significantly.
* Consumption of alcohol or smoking significantly.
* Taking anorexigenic or other weight-loss drugs (Xenical)
* Pregnant or breastfeeding
* Have polycystic ovary syndrome,
* Kidney failure
* Hypothyroidism,
* Cancer,
* Anxiety or depression

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Reduction in the prevalence of metabolic syndrome (obesity, diabetes, hypertension, dyslipidemia) | 24 weeks
  To first week(basal), 12 weeks after recruiting (intermediate) and 24 weeks after recruiting (final evaluation)

SECONDARY OUTCOMES:
Reduction of hyperglycemia | 24 weeks
  To first week(basal), 12 weeks after recruiting (intermediate) and 24 weeks after recruiting (final evaluation)
Weight loss | 24 weeks
  To first week(basal), 12 weeks after recruiting (intermediate) and 24 weeks after recruiting (final evaluation)
Reduction of high blood pressure | 24 weeks
  To first week(basal), 12 weeks after recruiting (intermediate) and 24 weeks after recruiting (final evaluation)
Reduction of hypercholesterolemia | 24 weeks
  To first week(basal), 12 weeks after recruiting (intermediate) and 24 weeks after recruiting (final evaluation)

CONTACTS AND LOCATIONS:
Overall Officials: Simón Barquera, PhD, Principal Investigator — Mexican National Institute of Public Health
Locations (1):
- Mexican National Institute of Public Health, Cuernavaca, Morelos, Mexico